CLINICAL TRIAL: NCT04559451
Title: Assessment of Remnant Liver Function in ALPPS by Gd-EOB-DTPA Enhanced MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTH-ALPPS
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Liver Function Failure; Liver Malignant Tumors
Keywords: Gd-EOB-DTPA Enhanced MRI; ALPPS; liver failure
MeSH Terms: conditions — Hepatic Insufficiency; Carcinoma, Hepatocellular; Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In order to further elucidate the molecular mechanism for the liver hypertrophy induced by the ALPPS, the blood sample and liver tissue sample before the first & second stage ALPPS operations will be collected under the permission of the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Insufficient future liver remnant (FLR), which may render post-hepatectomy liver failure, is one of the major obstacles for performing liver resection for patients with liver malignants. Associating liver partition and portal vein ligation (ALPPS) was introduced to induce rapid and extensive liver hypertrophy, which offers the opportunity for removing the liver malignancy in the second stage operation for patients with insufficient FLR at their first stage operation. Feasibility of the second stage of ALPPS has been assessed mostly on the basis of laboratory parameters and volumetry by the 3D reconstruction of CT. Meanwhile, part of the patients who underwent the second stage ALPPS still experienced postoperative liver failure, even in patients with sufficient FLR volume. In other words, this volumetric increase may not reflect the increase of liver function. And the laboratory parameters can only partly reflect the global liver function but not the regional liver function. Therefore, the combination of volumetric and global liver function tests might be unsuitable for predicting FLR function after first stage ALPPS because function is distributed unequally between left and right liver lobe. The Gd-EOB-DTPA-enhanced liver MRI, which has remarkable potential to evaluate regional liver function and could therefore be an ideal diagnostic test for performing volumetric and functional measurement after the first stage ALPPS in one examination. Thus we performed this clinical trial in order to evaluate the efficacy of Gd-EOB-DTPA-enhanced liver MRI in evaluating the FLR liver function after the first stage ALPPS.

DETAILED DESCRIPTION:
The clinical data and follow up information of the patients who underwent laparoscopic ALPPS in Department of General Surgery, Peking University Third Hospital were collected. The indication for the performance of the first and second ALPPS was evaluated by multi-disciplinary team (MDT). The liver function evaluation indexes of Gd-EOB-DTPA Enhanced liver MRI such as RE (Relative enhancement of the liver)=（SI20min-SIunenhanced）/ SIunenhanced and other related indexes were calculated. SI referred to signal intensity. SI20 min referred to the signal intensity in the hepatocyte phase (20 min after the injection). The relationship between the indexes and postoperative liver failure as well as other complications were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* future liver remnant volume <30%;
* indocyanine green clearance (ICG) rate <20% at 15 minutes;
* Child A liver function, serum platelet count > 50×109/L;
* good general condition.

Exclusion Criteria:

* complete right portal vein thrombosis;
* serum platelet count < 50×109/L;
* clinical signs of portal hypertension such as ascites, and/or intra-abdominal varices.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent ALPPS in Department of General Surgery, Peking University Third Hospital were collected. The indication for the performance of ALPPS were evaluated by multi-disciplinary team (MDT).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative liver function failure | Within 90 days after the operation
  The "50-50 criteria" was applied to assess post-treatment liver failure, which considers the increased total bilirubin level (>50 umol/L) and decreased PTA (<50%) on postoperative day 5.

SECONDARY OUTCOMES:
Postoperative morbidities and mortalities | Within 90 days after the operation
  Postoperative morbidities and mortalities were graded according to the Clavien classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China